CLINICAL TRIAL: NCT05605392
Title: Live Better at Home (Navarra): an Interventional Study
Brief Title: Live Better at Home, Navarra ( VMNav )
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Spanish Society of Geriatrics and Gerontology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VMCNav1.0
Record Dates: First submitted 2022-10-24; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Geriatrics; Institutionalization
Keywords: Older people; Deinstitutionalization; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deinstitutionalization (Experimental)
  Interventions: Other: Deinstitutionalization process

INTERVENTIONS:
Other: Deinstitutionalization process — Phase 1: Comprehensive geriatric assessment to evaluate who might be a candidate for deinstitutionalization.
  Phase 2: Intervention:
  1. Support plan: design a plan agreed upon with the participant to provide resources to the person's needs and which guarantees support during the transition and beyond.
  2. Transition process: progressive withdrawal of support in the institution and implementation of support and adaptation in the community, with different types of accommodation depending on the needs and preferences of each participant. Coordination with primary care teams, social services, and other community resources.
  3. Case follow-up and gradual withdrawal of the project team. If the process does not go as the person expects, or difficulties are encountered that cannot be resolved, the participant will have the option and choice, if desired, to return to the residence at any time during the process.

SUMMARY:
Alternatives to institutionalization with adapted housing and community supports may allow institutionalized people who so desire to be deinstitutionalized and continue their life in the community. This transition can fulfill the wishes of these people and may improve the quality of their life and functionality.

DETAILED DESCRIPTION:
Many older adults want to stay and be cared for at home, living in the community. However, long-term care facilities are increasingly becoming places where people live until death. Admissions are often conditioned by the characteristics of the support network rather than by the individual's clinical condition or dependency level. In addition, persistent problems around the cost and quality of housing with a lack of sufficient adapted housing and sheltered housing and inequalities in the distribution of social resources often limit the consolidation of personalized care and support planning.

Under this pretext, and if many people want to live at home for the rest of their lives, our research group aims to offer the possibility to nursing home residents from two nursing homes in Navarra of returning to the community by means of case management methodology and accommodation support. This completely innovative study aims to provide data to help the design and implementation of future studies addressed in this field.

The study consists of two stages:

1. A cross-sectional observational stage for the assessment. Objectives: Quantify the proportion of people who could return safely and quantify the proportion of people who would like to live in the community.
2. An analysis of factors related to the deinstitutionalization process and an intervention stage. Objective: assess the feasibility of this tailored intervention through case management methodology and study the impact of a deinstitutionalization process on participants for whom the transition is achieved.

In addition, this study will be accompanied by a sub-study with a pseudo-qualitative approach. The main objective of this part is to characterize the discourses associated with the willingness to return to the community and the deinstitutionalization process and to identify which evaluative elements concur (barriers and facilitators) and are prioritized in decision-making about a possible deinstitutionalization process. Qualitative research is needed for complex interventions to explore the obstacles and facilitators and to understand the intervention's components.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* To have a place within the recruitment period for an indefinite period of time in one of the participating centers.

Phase 2:

* To express willingness to be deinstitutionalized and return to community.
* To obtain a favorable report in phase 1 from the project team on the feasibility and safety of returning to community.

Exclusion Criteria:

* Refusal to sign the informed consent form by the resident or, failing that, by the legal representative.
* The existence of a judicial authorization for involuntary admission of the resident to the residential facility.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-03-28 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life. | Every three months after signing the personalized support plan (baseline) up to 15 months
  Assessed by Fumat Scale. Standard score (M= 10; Standard deviation (SD)= 3) of each quality of life dimension, percentiles, and quality of life Index

SECONDARY OUTCOMES:
Functional capacity. | Every 3 months up to 15 months
  Assessed by the Barthel Index. The scoring rate is from 0 (total dependency)- 100 (slight dependency)
Frailty. | Every 3 months up to 15 months
  Assessed by the Frail-VIG Index. The scoring range is from 0 (no frailty)- 25 (advanced frailty)
Cognitive status. | Every 3 months up to 15 months
  Assessed by the mini-mental test. The scoring range is from 0 (severe cognitive impairment) to 30 (no cognitive impairment)
Change on performance activities of daily living. | Every 3 months up to 15 months
  Assessed by BELS (Basic Everyday Living Skills). It consists of two scales: one to evaluate the opportunity to performance (from 0- no opportunity to 2- total opportunity) and the other for the real performance of activities (from 0- no performance of any activity- to 4- normal level of performance).
Physical Activity | Every 3 months up to 15 months
  Assessed by IPAQ questionnaire. The classification ranges from a low level of physical activity to high level of physical activity.
Depression | Every 3 months up to 15 months
  Assessed by Yesavage Geriatric Depression Scale. The scoring range is from 0 (no depression) - 10 (high depression)
Loneliness | Every 3 months up to 15 months
  Assessed by ESTE Scale. The scoring range is from 0 (low degree)- 30 (high degree)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Augusto García Navarro, Principal Investigator — Spanish Society of Geriatrics and Gerontology
Locations (2):
- Spain (2):
  - Residencia Santo Domingo, Estella-Lizarra, Navarre
  - Residencia El Vergel, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: Yes
All collected data will result in some publications
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Access criteria will be made on demand

REFERENCES:
- [Derived] Roncal-Belzunce V, Atares L, Escalada G, Minobes-Molina E, Pamies-Tejedor S, Carcavilla-Gonzalez N, Garcia-Navarro JA. First steps towards the deinstitutionalization of older adults: A protocol for the implementation of a complex intervention. Rev Esp Geriatr Gerontol. 2024 Mar-Apr;59(2):101453. doi: 10.1016/j.regg.2023.101453. Epub 2023 Dec 15. PMID 38103438